CLINICAL TRIAL: NCT06419309
Title: Comparison of the Effect of Gluten-Free-Lactose-Free / Aronia Melanocarpa Supplemented Diet on Leptin, Ghrelin Levels and Inflammatory Status in Patients With Hashimoto Thyroiditis
Brief Title: Comparison of the Effect of Gluten-Free-Lactose-Free / Aronia Melanocarpa Supplemented Diet in Patients With Hashimoto's Thyroiditis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUSBFBVDBE001
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Hashimoto Thyroiditis
MeSH Terms: conditions — Hashimoto Disease | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gluten- lactose free diet (Experimental): People will be given a healthy diet by eliminating gluten-free lactose-containing foods from their diet. It will continue for 8 weeks.
  Interventions: Other: Dietary intervention
- Aronia Melanocarpa added and Gluten- lactose free diet (Experimental): In addition to a healthy diet, people will be given aronia melanocarpa fruit juice daily (high in anthocyanins, 69.24 mg/100 mL cyanidin-3-glucoside) and a gluten-free-lactose-free diet.It will continue for 8 weeks.
  Interventions: Other: Dietary intervention
- Aronia Melanocarpa added diet (Experimental): People will be given aronia melanocarpa fruit juice daily (high in anthocyanins, 69.24 mg/100 mL cyanidin-3-glucoside).It will continue for 8 weeks.
  Interventions: Other: Dietary intervention
- Healthy eating group (Experimental): Healthy diet patterns with an average macronutrient content of 10-20% protein, 20-35% fat and 45-60% carbohydrate will be followed for 8 weeks.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Four different dietary interventions are planned.
  * Gluten-free, lactose-free diet,
  * Diet enriched with Aronia Melanocarpa,
  * Gluten-free, lactose-free and enriched with Aronia Melanocarpa diet,
  * Healthy diet

SUMMARY:
Hashimoto's thyroiditis (HT) is the most common cause of chronic hypothyroidism in areas with sufficient iodine, stemming from an autoimmune response against thyroid peroxidase and/or thyroglobulin. It is the most prevalent autoimmune thyroid disease and a leading cause of overall hypothyroidism. Even when they reach euthyroidism, 82% of treated women with HT still have excess body weight, and 35% of them are obese. Thyroid dysfunction can affect the function of adipose tissue and lead to metabolic disturbances. Leptin can stimulate thyroid-stimulating hormone secretion, while thyroid-stimulating hormone can influence leptin release from adipose tissue. Additionally, HT patients often exhibit high levels of C-reactive protein and interleukin-6, suggesting an association between increased thyroid-stimulating hormone levels and the inflammatory process, which may contribute to comorbid disease risk in individuals with HT. Nutrition can serve as a complementary treatment for HT by affecting thyroid functions and having anti-inflammatory properties. Dietary interventions may involve eliminating gluten, lactose, or certain food components, or focusing on an anti-inflammatory dietary pattern while preventing nutritional deficiencies. Therefore, this study is a randomized controlled, single-blind trial designed to evaluate the effects of a gluten-free, lactose-free diet and a diet enriched with Aronia Melanocarpa, both individually and in combination, as well as healthy dietary protocols, on autoantibody levels, leptin, ghrelin, oxidative response, and weight loss in patients with Hashimoto's thyroiditis. The study aims to recruit a minimum of 80 participants aged 18-65 years, diagnosed with Hashimoto's thyroiditis at Istanbul Medical Faculty Hospital. In the initial face-to-face interview, participants will provide sociodemographic information, dietary habits, anthropometric measurements, and dietary intake records through a questionnaire. The study involves the inclusion of Aronia Melanocarpa in the diet (high anthocyanin content, 69.24 mg/100 ml), a gluten-free and lactose-free diet, both interventions being applied together, and the application of only healthy nutrition protocols to patients over an 8-week period, with serum assessments of thyroid-stimulating hormon, free T4, free T3, anti-thyroid peroxidase, anti-Tg, interleukin-6,anti tumor necrosis factor alpha, C-reactive protein and leptin-ghrelin levels at the beginning and end of the study. The goal is to create recommendations for patients, improve their quality of life, and establish sustainable nutritional interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Hashimoto's thyroiditis by a doctor,
* Being a female individual between the ages of 18-65,
* Not being diagnosed with any chronic disease that would negatively affect functioning other than Hashimoto's thyroid,
* Not having used selenium and iodine supplements in the last month,
* Individuals should not lose more than 4 kg of weight in the last month,
* Not having been on a strict elimination diet for more than 4 months in the last year,
* Not having applied any nutritional intervention during the last three months before the study.

Exclusion Criteria:

* Pregnant or breastfeeding mother,
* Individuals with chronic diseases,
* Individuals allergic to red fruits

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the prevalence of the disease is high in female individuals, it will be conducted with female individuals.
Enrollment: 80 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Effect of diet on weight loss | Start and end of study (8 weeks)
  The effect of diets on weight loss will be evaluated. Body composition analyzes of individuals (body weight (kg), body fat ratio (%), body water ratio (%), visceral fat ratio) will be performed using handheld device.
Effect of diet on hormone level | Start and end of study (8 weeks)
  The effects of diets on leptin and ghrelin levels will be examined with venous blood samples.
Effect of diet on inflammatory parameters | Start and end of study (8 weeks)
  To evaluate oxidative stress parameters, two 5 mL venous blood samples will be taken from each patient in yellow tubes after an overnight fast of at least eight hours between 08:00 and 09:00 in the morning.
  The blood sample will be kept at room temperature for 10-20 minutes and after being centrifuged at 2000-3000 rpm for 20 minutes, it will be transferred to Eppendorf tubes with the help of a sterile pipette and will be stored in 2 separate refrigerators at -20 °C.
  IL-6, TNF-alpha, CRP levels will be measured with commercial kits, following the company protocol.

SECONDARY OUTCOMES:
Effect of diet on routine hashimoto thyroid parameters | Start and end of study (8 weeks)
  Thyroid Stimulating Hormone, free thyroxine, free triiodothyronine, thyroid peroxidase antibodies and anti-thyroglobulin biochemical parameters of the participants will be requested by the doctor with institutional permission and patient approval.

CONTACTS AND LOCATIONS:
Overall Officials: Berrak Basturk, Lecturer, Principal Investigator — Halic University; Zeynep Ozerson, Assoc. prof., Study Director — Halic University; Ayse Kubat Uzum, Profesor, Study Director — Istanbul University; Melike Cevikdizici, Nurse, Study Director — Istanbul University; Yusuf Celik, Profesor, Study Director — Biruni University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)